CLINICAL TRIAL: NCT04998474
Title: A Phase II Trial of Personalized Tumor Neoantigen Based Vaccine FRAME-001 for Advanced Non-Small Cell Lung Cancer
Brief Title: FRAME-001 Personalized Vaccine in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Frame Pharmaceuticals B.V. (Industry)
Collaborators: Erasmus Medical Center (Other); The Netherlands Cancer Institute (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRAME-001
Record Dates: First submitted 2021-07-01; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FRAME-001 personalized vaccine (Experimental): Prospective, single arm, multi center, open-label, phase II clinical trial.
  Patients will receive personalized peptide vaccine FRAME-001 based on frame-shift mutations (Frames) detected by Whole Genome Sequencing (WGS)/Ribonucleic Acid sequencing (RNAseq) in a tumor biopsy. FRAME-001 vaccine will be administered in four sequential cycles at 3-week interval (Q3W), along standard maintenance monotherapy of pembrolizumab (administration Q3W or Q6W). Each cycle will be consisting of up to four subcutaneous injections at up to four different sites in the upper and lower limbs.
  Interventions: Biological: FRAME-001 personalized vaccine

INTERVENTIONS:
Biological: FRAME-001 personalized vaccine — Patients will receive personalized peptide vaccine FRAME-001 based on frame-shift mutations (Frames) detected by Whole Genome Sequencing (WGS)/Ribonucleic Acid sequencing (RNAseq) in a tumor biopsy. FRAME-001 vaccine will be administered in four sequential cycles at 3-week interval (Q3W), along standard maintenance monotherapy of pembrolizumab (administration Q3W or Q6W). Each cycle will be consisting of up to four subcutaneous injections at up to four different sites in the upper and lower limbs.

SUMMARY:
Despite encouraging results of programmed cell death protein -1 (PD-1) immune checkpoint inhibitor treatment combined with chemotherapy in advanced non-small cell lung cancer (NSCLC), only the minority of approximately 20% of patients derive durable clinical benefit from such treatment. Patients with stable disease (SD) after four cycles of treatment with PD-1 inhibitor pembrolizumab monotherapy or in combination with chemotherapy (standard of care in advanced NSCLC in the Netherlands) have a low probability of still acquiring a complete response (CR) or durable disease control to such treatment and no other curative standard treatment options are available, emphasizing the need for novel therapeutic approaches. Tumor-specific neopeptides resulting from frameshift mutations in tumor cells, so-called Frames, present potentially potent targets for the immune system and can be utilized in therapeutic anti-cancer vaccination with the intention to synergize in their effect with immune chckpoint inhibitors. Frames are prevalent in NSCLC patients, with 95% of lung tumors harboring one or more Frames. The entire collection of Frames expressed by a tumor is referred to as the Framome. Vaccination against strongly antigenic neopeptides present in a patient's tumor furnishes a perspective of enhancing the therapeutic effect of the immune checkpoint inhibition in NSCLC with expected limited additional toxicities. The current clinical trial is designed to determine immune response, safety, and clinical response of personalized vaccine FRAME-001 based on a patient's Framome and selection of Frame peptides in advanced NSCLC cancer patients after standard first line treatment consisting of immune checkpoint inhibitor pembrolizumab as monotherapy or combined with chemotherapy (carboplatin/cisplatin and pemetrexed/paclitaxel), and who attained SD after four cycles of such therapy. The personalized FRAME-001 vaccine will be administered during maintenance phase of treatment with pembrolizumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically and radiologically confirmed advanced squamous or non-squamous NSCLC with SD after four cycles of treatment with pembrolizumab as monotherapy or in combination with chemotherapy (carboplatin/cisplatin and pemetrexed/paclitaxel) and suitable for maintenance treatment with pembrolizumab monotherapy.
* Patient Framome identification and characterization with demonstrated expressed at least three frameshift mutations (Frames) with combined ³100 amino acids (preferably more than 100 amino acids) completed as part of molecular pre-screening.
* Eastern Cooperative Oncology Group (ECOG) £1.
* An expected survival of at least 3 months.
* Presence of tumor lesion(s) suitable for biopsy and radiological assessment as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
* Written informed consent according to International Conference on Harmonisation (ICH)-Good Clinical Practice (GCP).

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Any active infection that might according to investigator interfere with FRAME-001 vaccination.
* Current use of systemic corticosteroids (or other immunosuppressive agents; >10mg daily prednisone equivalent). Inhaled, intranasal or topical and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted.
* Live vaccine within 30 days prior to first dose of FRAME-001.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
FRAME-001-specific immune responses in peripheral blood after administration of FRAME-001 | Week 7, 10, 13, 16, 19 and week 49
  Antigen-specific immune responses in peripheral blood to one or more Frame peptides following application of a personalized FRAME-001 vaccine, based on a positive outcome in one or more of the following assays:
  1. 4-Day interferon gamma (IFNg) enzyme-linked immunospot (ELISpot) assay.
  2. IFNg, tumor necrosis factor alpha (TNFa), and/or interleukin-2 (IL-2) producing CD4+ and/or CD8+ T cells determined in intracellular cytokine staining assay.
  3. Specific cytokine production as measured by Th1/Th2 cytokine bead array in culture supernatants.

SECONDARY OUTCOMES:
The number of adverse events (AEs) according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. | Up to week 22
  Assessment of safety and tolerability of FRAME-001
Evaluation of clinical anti-tumor response and survival after treatment with FRAME-001 | Through study completion, an average of 2 years
  Tumor response and tumor response duration according to Response Evaluation Criteria in Solid Tumors (RECIST) v.1.1 criteria. And progression-free survival (PFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Bob Löwenberg, MD, Study Chair — Frame Pharmaceuticals B.V.; J.G.J.V. Aerts, MD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam
  - University Medical Center Groningen, Groningen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No